CLINICAL TRIAL: NCT00485355
Title: A Prospective Randomized Trial Comparing Conventional vs. Robotic Assisted Laparoscopic Hysterectomy
Brief Title: Study Comparing Conventional vs. Robotic-assisted Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-150
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2013-08

CONDITIONS: Uterine Fibroids, Menorrhagia, Endometriosis
Keywords: hysterectomy; Laparoscopy; robotics
MeSH Terms: conditions — Leiomyoma; Menorrhagia; Endometriosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Conventional Laparoscopic Hysterectomy
  Interventions: Procedure: conventional laparoscopic hysterectomy
- 2 (Active Comparator): Robotic Assisted Laparoscopic Hysterectomy
  Interventions: Procedure: robotic assisted laparoscopic hysterectomy

INTERVENTIONS:
Procedure: conventional laparoscopic hysterectomy — Total laparoscopic hysterectomy
  Arms: 1
Procedure: robotic assisted laparoscopic hysterectomy — Robotic assisted laparoscopic hysterectomy with DaVinci robot
  Arms: 2

SUMMARY:
The purpose of this study is to compare two ways of performing laparoscopic hysterectomy - robotic-assisted vs. conventional laparoscopy.

DETAILED DESCRIPTION:
Compared to abdominal hysterectomy, the advantages of laparoscopic hysterectomy are decreased postoperative intravenous analgesia requirements, shorter length of hospital stay, quicker return to work and daily activities. Longer operating times have been shown to be offset by shorter hospital stays, with similar hospital costs overall. Compared to abdominal hysterectomy, laparoscopic hysterectomy is associated with less blood loss, fewer abdominal wall infections, or febrile episodes. The increased visualization allows for concomitant evaluation and excision of adhesions or endometriosis, as well as facilitating oophorectomy.

Robotic systems were developed in order to facilitate laparoscopy by more ergonomic movements that are easier to perform and more precise. The da Vinci Surgical System (Intuitive Surgical Inc., Sunnyvale, CA, USA) has endowrist instruments that have seven degrees of movement and mimic the human wrist. It can also filter out tremors and other unintentional hand motions that may result from prolonged holding of instruments. The surgeon seated at a console commands the laparoscope and two laparoscopic surgical instruments.

In the literature, several case series have described the use of robotic-assisted hysterectomy. Two of these series included patients that were undergoing surgery for suspected malignancy, and hence has a different patient population that we are going to enroll.Overall these studies have demonstrated the feasibility of using robot-enhanced technology in order to perform hysterectomy in series of approximately 10-20 patients, with a similar rate of complications compared to classical laparoscopy.

The objective of this study is to conduct a prospective randomized controlled trial of robotic assisted versus traditional hysterectomy in the treatment of patients who have benign indications for hysterectomy, e.g. menorrhagia, symptomatic fibroid uteri, etc. Our primary outcome is operative time from incision to either closure or, in the case of concomitant prolapse or incontinence procedures, the completion of the hysterectomy portion of the case, i.e. closure of vaginal cuff and achievement of hemostasis from the hysterectomy. Secondary outcomes include intra-operative, peri-operative, and post-operative complications; post-operative patient outcomes as measured by the Short Form 36 (SF-36) questionnaire. Patient scores on this questionnaire before and after surgery can be used to calculate the quality adjusted life years (QALYs), which can then be used in the cost utility analysis. Patients' overall narcotic use and quality of life will also be assessed after surgery with diaries at different intervals. The diaries will consist of a daily narcotic/pain medication diary, a weekly assessment of return to normal activity, and assessments at 2, 4, and 6 weeks of surgical pain and ability to perform functional activities.

ELIGIBILITY:
Inclusion Criteria:

* women who are 18 years of age or greater who are to undergo laparoscopic hysterectomy for benign indications. Other concomitant laparoscopic or anti-incontinence procedures (e.g., excision of endometriosis or mid-urethral sling procedures) will be performed at the primary surgeon's discretion.

Exclusion Criteria:

* suspected malignancy, medical illness precluding laparoscopy, inability to give informed consent, morbid obesity (BMI>40), or need for concomitant bowel resection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Operative time from incision to either closure or, in the case of concomitant prolapse or incontinence procedures, the completion of the hysterectomy portion of the case, i.e. closure of vaginal cuff and achievement of hemostasis from the hysterectomy. | Intra-operative time

SECONDARY OUTCOMES:
Peri-operative complications; comparison of costs; qualify of life issues; post-operative pain and narcotic use; return to normal activity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie FR Paraiso, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Result] Paraiso MF, Ridgeway B, Park AJ, Jelovsek JE, Barber MD, Falcone T, Einarsson JI. A randomized trial comparing conventional and robotically assisted total laparoscopic hysterectomy. Am J Obstet Gynecol. 2013 May;208(5):368.e1-7. doi: 10.1016/j.ajog.2013.02.008. Epub 2013 Feb 8. PMID 23395927